CLINICAL TRIAL: NCT02262754
Title: A Randomized, Double Blind, Placebo- And Active-controlled, 4 Week, Multi-center, Parallel Group Study Assessing The Analgesic Effect, Safety And Tolerability Of Pf-06372865 In Subjects With Chronic Low Back Pain Using Naproxen As Positive Control
Brief Title: PF-06372865 In Subjects With Chronic Low Back Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B7431006
Record Dates: First submitted 2014-10-09; First posted 2014-10-13 (Estimated); Results first posted 2017-01-04 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Low Back Pain
MeSH Terms: interventions — PF-06372865; Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- PF-06372865 (Experimental): Daily BID dosing for 4 weeks
  Interventions: Drug: PF-06372865
- Placebo (Placebo Comparator): Daily BID dosing for 4 weeks
  Interventions: Drug: Placebo
- Naproxen (Active Comparator): Daily BID dosing for 4 weeks
  Interventions: Drug: Naproxen

INTERVENTIONS:
Drug: PF-06372865 — Dose level 1 daily dosing BID for 1 week followed by dose level 2 daily BID for 3 weeks
  Arms: PF-06372865
Drug: Placebo — Placebo for PF-06372865 and placebo for naproxen daily
  Arms: Placebo
Drug: Naproxen — 500 mg BID for 4 weeks
  Arms: Naproxen

SUMMARY:
PF-06372865 In Subjects With Chronic Low Back Pain

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2014-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (46):
- United States (46):
  - Agave Clinical Research, LLC, Mesa, Arizona
  - Arizona Research Center, Inc., Phoenix, Arizona
  - Global Research, Anaheim, California
  - Neuro-Pain Medical Center, Fresno, California
  - Providence Clinical Research, North Hollywood, California
  - Elite Clinical Trials, Incorporate, Wildomar, California
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Avail Clinical Research, LLC, DeLand, Florida
  - S&W Clinical Research, Fort Lauderdale, Florida
  - Florida Research Network, LLC, Gainesville, Florida
  - Broward Research Group, Hollywood, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Compass Research, LLC, Orlando, Florida
  - Pines Clinical Research Inc., Pembroke Pines, Florida
  - Accord Clinical Research, LLC, Port Orange, Florida
  - Arthritis & Rheumatic Care Center, South Miami, Florida
  - Miami Research Associates, South Miami, Florida
  - Better Health Clinical Research, Inc., Atlanta, Georgia
  - River Birch Research Alliance, LLC, Blue Ridge, Georgia
  - Family Medicine center, Columbus, Georgia
  - Columbus Regional Research Institute, Columbus, Georgia
  - Drug Studies America, Marietta, Georgia
  - Better Health Clinical Research, Inc./Georgia Pain & Spine Care, Inc., Newnan, Georgia
  - Better Health Clinical Research, Inc., Newnan, Georgia
  - Southeast Regional Research Group, Savannah, Georgia
  - North Georgia Clinical Research, Woodstock, Georgia
  - North Georgia Internal medicine, Woodstock, Georgia
  - Chicago Anesthesia Associates, Chicago, Illinois
  - Centex Studies, Inc, Lake Charles, Louisiana
  - Boston Clinical Trials, Boston, Massachusetts
  - ActivMed Practices & Research, Inc., Methuen, Massachusetts
  - CRC of Jackson, Jackson, Mississippi
  - Physician's Surgery Center, Jackson, Mississippi
  - Drug Trials America, Hartsdale, New York
  - AAIR Research Center, Rochester, New York
  - Wake Internal Medicine Consultants, Inc., Raleigh, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Summit Research Network (Oregon), Inc., Portland, Oregon
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Clinical Trial Network, Houston, Texas
  - Lee Medical Associates, PA, San Antonio, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - National Clinical Research - Norfolk, Inc., Norfolk, Virginia
  - Summit Research Network (Seattle) LLC, Seattle, Washington

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7431006&StudyName=A%20Randomized%2C%20Double%20Blind%2C%20Placebo-%20And%20Active-controlled%2C%204%20Week%2C%20Multi-center%2C%20Parallel%20Group%20Study%20Assessing%20The%20Analgesic%20Effect%2C%20Safety%20And%20Tolerability%20Of%20Pf-06372865%20In%20Subjects%20With%20Chronic%20Low%20Back%20Pain%20Using%20Naproxen%20As%20Positive%20Control

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebo matched to PF-06372865 tablets along with Naproxen 500 milligram (mg) tablets orally, twice daily for four weeks.
- PF-06372865: Participants received PF-06372865 2.5 mg tablets along with placebo matched to Naproxen tablets orally, twice daily for one week followed by PF-06372865 7.5 mg tablets along with placebo matched to Naproxen tablets orally, twice daily for three weeks.
- Naproxen: Participants received Naproxen 500 mg tablets along with placebo matched to PF-06372865 tablets orally, twice daily for four weeks.
Period: Overall Study
Arm/Group | Placebo | PF-06372865 | Naproxen
Started | 74 | 74 | 74
Completed | 58 | 65 | 65
Not Completed | 16 | 9 | 9
Not completed — Adverse Event | 3 | 4 | 0
Not completed — Lack of Efficacy | 2 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — No longer meets eligibility criteria | 0 | 1 | 0
Not completed — Study terminated by sponsor | 5 | 4 | 4
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Other | 4 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all participants randomized and who had received at least 1 dose of randomized treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | PF-06372865 | Naproxen | Total
Number analyzed (Participants) | 74 | 74 | 74 | 222
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (12.1) | 49.7 (13.8) | 51.6 (13.1) | 50.8 (12.9)
Gender [Count of Participants; unit: Participants]
  FEMALE | 38 | 39 | 37 | 114
  MALE | 36 | 35 | 37 | 108

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Daily Low Back Pain Intensity (LBPI) Score as Measured by an 11-point Numeric Rating Scale (NRS) at Week 4
Description: Daily average low back pain was assessed on an 11-point numeric rating scale (NRS). Participants described their average low back pain during the past 24 hours on a scale ranging from 0 (no pain) to 10 (worst possible pain), where higher scores indicate higher pain. Baseline value was calculated as the mean of the scores over the last 7 days in the placebo run-in period, prior to randomization. Post-baseline weekly scores were calculated based on the mean of the scores over the 7 days prior to and including the day at the end of the corresponding week.
Time Frame: Baseline, Week 4
Population: FAS included all participants randomized and who had received at least 1 dose of randomized treatment.
Measure: Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | PF-06372865 | Naproxen
Number analyzed (Participants) | 74 | 74 | 74
units on a scale | -1.19 (1.351) [-1.50 to -0.89] | -1.03 (1.091) [-1.35 to -0.71] | -1.45 (1.401) [-1.77 to -1.14]
Statistical Analysis 1: Comparison: Placebo vs PF-06372865; An analysis of covariance (ANCOVA) model within an outlier robust Bayesian framework was applied. Baseline was included as a fixed effect. An informative N (-2.36, 0.542^2) prior for the placebo effect was assumed. Non informative prior distributions were assumed for the rest of the model parameters. A last observation carried forward (LOCF) was used for missing data; Test type: Superiority or Other; Mean Difference (PF-06372865-Placebo) = 0.16, 90% CI 2-sided [-0.28 to 0.60]
Statistical Analysis 2: Comparison: PF-06372865 vs Naproxen; An ANCOVA model within an outlier robust Bayesian framework was applied. Baseline was included as a fixed effect. An informative N (-2.36, 0.542^2) prior for the placebo effect was assumed. Non informative prior distributions were assumed for the rest of the model parameters. A last observation carried forward LOCF was used for missing data; Test type: Superiority or Other; Mean Difference (PF-06372865-Naproxen) = 0.42, 90% CI 2-sided [-0.02 to 0.87]
Statistical Analysis 3: Comparison: Placebo vs Naproxen; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; Mean Difference (Naproxen-Placebo) = -0.26, 90% CI 2-sided [-0.70 to 0.18]

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. The SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death, initial or prolonged inpatient hospitalization, life-threatening experience (immediate risk of dying), persistent or significant disability or incapacity, congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. AEs included both serious and non-serious adverse events.
Time Frame: Baseline up to 28 days after the last dose of study treatment (Day 56)
Population: Safety analysis set included all participants who received at least 1 dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-06372865 | Naproxen
Number analyzed (Participants) | 74 | 74 | 74
participants
  AEs | 26 (1.351) [-1.50 to -0.89] | 34 (1.091) [-1.35 to -0.71] | 28 (1.401) [-1.77 to -1.14]
  SAEs | 1 | 1 | 2

3. Primary Outcome: Number of Participants With Laboratory Abnormalities
Description: Abnormality criteria included: hemoglobin, hematocrit and red blood cells (RBCs) (less than [<] 0.8*lower limit of normal [LLN]); white blood cells (WBC) (<0.6*LLN, greater than [>] 1.5*upper limit of normal [ULN]); MCV, MCH, MCHC (<0.9*LLN, >1.1*ULN); platelets (<0.5*LLN>, >1.75*ULN); neutrophils, lymphocytes(<0.8*LLN, >1.2*ULN); eosinophils, basophils, monocytes (>1.2*ULN); total bilirubin (>1.5*ULN); aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase (>3*ULN); total protein, albumin (<0.8*LLN, >1.2*ULN); creatinine, blood urea nitrogen (>1.3*ULN); glucose (<0.6*LLN, >1.5*ULN); uric acid (>1.2*ULN); sodium, potassium, chloride, calcium, bicarbonate (<0.9*LLN, >1.1*ULN); urine pH (<4.5, >8); qualitative urine glucose, ketones, protein, blood values (greater than or equal to [>=] 1) in urine dipstick test; urine RBC, WBC (>=20); hyaline casts (>1), bacteria (>20).
Time Frame: Baseline up to 28 days after the last dose of study treatment (Day 56)
Population: Safety analysis set included all participants who received at least 1 dose of study treatment. Here, "number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-06372865 | Naproxen
Number analyzed (Participants) | 73 | 74 | 74
participants | 26 | 44 | 41

4. Primary Outcome: Number of Participants With Vital Sign Abnormalities
Description: Participants who met the criteria for abnormal findings in vital signs data were reported. Criteria for abnormalities in vital signs: supine systolic blood pressure (SBP) <90 millimeter of mercury (mmHg), supine diastolic BP (DBP) <50 mmHg, supine pulse rate <40 beats per minute (bpm) or >120 bpm. Maximum increase or decrease from baseline in supine SBP >=30 mmHg and maximum increase or decrease from baseline in supine DBP >=20 mmHg.
Time Frame: Baseline up to Follow-up (44 days)
Population: Safety analysis set included all participants who received at least 1 dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-06372865 | Naproxen
Number analyzed (Participants) | 74 | 74 | 74
participants
  Supine SBP: <90 mmHg | 0 (1.351) [-1.50 to -0.89] | 1 (1.091) [-1.35 to -0.71] | 0 (1.401) [-1.77 to -1.14]
  Supine DBP: <50 mmHg | 0 | 1 | 0
  Supine pulse rate: <40 bpm | 0 | 0 | 0
  Supine pulse rate: >120 bpm | 0 | 0 | 0
  Maximum increase in Supine SBP: >=30 mmHg | 5 | 0 | 1
  Maximum increase in Supine DBP: >=20 mmHg | 6 | 3 | 4
  Maximum decrease in Supine SBP: >=30 mmHg | 1 | 6 | 4
  Maximum decrease in Supine DBP: >=20 mmHg | 3 | 9 | 3

5. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities
Description: Participants with abnormal ECG findings were reported. Criteria for potential clinical concern in ECG parameters: maximum (max.) PR interval of >=300 milliseconds (msec), maximum QRS interval >=140 msec, maximum QTCF interval (Fridericia's Correction) of 450 to <480 msec, 480 to <500 msec and >=500 msec, maximum of >=25 percent (%) increase from baseline (IFB) value of >200 msec and >=50% for baseline value of less than or equal to (<=) 200 msec for PR interval, maximum increase from baseline of >=50% for QRS interval, maximum increase from baseline of >=30 msec to <60 msec and maximum increase from baseline of >60 msec in QTCF interval (Fridericia's Correction).
Time Frame: Baseline up to Follow-up (44 days)
Population: Safety analysis set included all participants who received at least 1 dose of study treatment. Here, "n" signifies the number of participants evaluable for the specific category.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-06372865 | Naproxen
Number analyzed (Participants) | 74 | 74 | 74
participants
  Max. PR Interval: >=300 msec (n=72, 74, 72) | 0 (1.351) [-1.50 to -0.89] | 0 (1.091) [-1.35 to -0.71] | 0 (1.401) [-1.77 to -1.14]
  Max. QRS Complex: >=140 msec (n=72, 74, 72) | 0 | 0 | 1
  Max. QTCF Interval: 450 to <480 msec (n=72,74,72) | 1 | 1 | 2
  Max. QTCF Interval: 480 to <500 msec (n=72,74,72) | 0 | 1 | 0
  Max. QTCF Interval: >=500 msec (n=72, 74, 72) | 0 | 0 | 0
  Max. PR Interval IFB: >=25 or 50% (n=72, 74, 71) | 1 | 0 | 0
  Max. QRS Complex IFB: >=50% (n=72, 74, 72) | 1 | 0 | 1
  Max. QTCF Interval IFB: 30 to<60 msec (n=72,74,72) | 3 | 4 | 0
  Max. QTCF Interval IFB: >=60 msec (n=72,74,72) | 3 | 1 | 0

6. Primary Outcome: Number of Participants With Categorical Scores on the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS (mapped to Columbia Classification Algorithm of Suicide Assessment [C-CASA]) is an interview-based rating scale to systematically assess suicidal ideation and suicidal behavior. C-SSRS assessed whether participant experienced following: completed suicide =1, suicide attempt =2 (response of "Yes" on "actual attempt"), preparatory acts toward imminent suicidal behavior =3 ("Yes" on "preparatory acts or behavior"), suicidal ideation =4 ("Yes" on "wish to be dead", "non-specific active suicidal thoughts", "active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent), any suicidal behavior or ideation, self-injurious behavior =7 ("Yes" on "Has participant engaged in non-suicidal self-injurious behavior").
Time Frame: Screening, Baseline, Week 1, 2, 3, 4
Population: Data was not collected for this outcome measure as per study team's decision, since it was a semi-structured interview and was difficult to pull accurate scores from it.
Arm/Group | Placebo | PF-06372865 | Naproxen
Number analyzed (Participants) | 0 | 0 | 0

7. Primary Outcome: Change From End of Treatment Visit in Physician's Withdrawal Checklist (PWC) Score at Follow-up Visit
Description: PWC is a 20 item physician rated interview to measure anxiolytic drug withdrawal-related signs and symptoms. Each individual item score ranges from 0 (not present) to 3 (severe), where higher scores = more affected condition. PWC total score range from 0 (not present) to 60 (severe), where higher score = more affected condition. Change: score at follow-up visit minus score at the end of treatment visit.
Time Frame: End of treatment (Day 30), follow-up (Day 44)
Population: Safety analysis set included all participants who received at least 1 dose of study treatment.
Measure: Least Squares Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | PF-06372865 | Naproxen
Number analyzed (Participants) | 74 | 74 | 74
units on a scale | -0.11 (1.351) [-0.49 to 0.28] | -0.34 (1.091) [-0.71 to 0.03] | 0.01 (1.401) [-0.36 to 0.38]
Statistical Analysis 1: Comparison: Placebo vs PF-06372865; The ANCOVA model included treatment as fixed effects; Test type: Superiority or Other; LS Mean Difference (PF-06372865-Placebo) = -0.23, 90% CI 2-sided [-0.76 to 0.30], Standard Error of Mean 0.32
Statistical Analysis 2: Comparison: Placebo vs Naproxen; The ANCOVA model included treatment as fixed effects; Test type: Superiority or Other; LS Mean Difference (Naproxen-Placebo) = 0.12, 90% CI 2-sided [-0.41 to 0.65], Standard Error of Mean 0.32
Statistical Analysis 3: Comparison: PF-06372865 vs Naproxen; The ANCOVA model included treatment as fixed effects; Test type: Superiority or Other; LS Mean Difference(PF-06372865-Naproxen) = -0.35, 90% CI 2-sided [-0.87 to 0.17], Standard Error of Mean 0.32

8. Secondary Outcome: Change From Baseline in Daily Low Back Pain Intensity (LBPI) as Measured by an 11-point Numeric Rating Scale (NRS) at Week 1, 2 3 and 4
Description: Average back pain was assessed with an 11-point NRS ranging from 0 (no pain) to 10 (worst possible pain), where higher scores indicated higher pain. Participants described their average low back pain during the past 24 hours by choosing the appropriate number from 0 to 10.
Time Frame: Baseline, Week 1, 2, 3, 4
Population: FAS included all participants randomized and who had received at least 1 dose of randomized treatment. Here, "n" signifies participants who were evaluable at the specified time point for each arm.
Measure: Least Squares Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | PF-06372865 | Naproxen
Number analyzed (Participants) | 74 | 74 | 74
units on a scale
  Change at week 1 (n= 74, 74, 74) | -0.50 (1.351) [-0.69 to -0.30] | -0.41 (1.091) [-0.61 to -0.22] | -0.70 (1.401) [-0.90 to -0.50]
  Change at week 2 (n= 65, 70, 72) | -0.93 [-1.21 to -0.65] | -0.98 [-1.25 to -0.70] | -1.17 [-1.44 to -0.90]
  Change at week 3 (n= 62, 69, 70) | -1.12 [-1.43 to -0.82] | -1.09 [-1.39 to -0.80] | -1.39 [-1.68 to -1.10]
  Change at week 4 (n= 59, 64, 66) | -1.22 [-1.56 to -0.87] | -1.14 [-1.48 to -0.81] | -1.58 [-1.91 to -1.25]
Statistical Analysis 1: Comparison: Placebo vs PF-06372865; Week 1: The mixed effect repeated measures model was used and included treatment, week, baseline, the week * treatment interaction, and the baseline * week interaction as fixed effects and week repeated within each participant as a repeated effect. Baseline was included as a covariate; Test type: Superiority or Other; LS Mean Difference (PF-06372865-Placebo) = 0.08, 90% CI 2-sided [-0.20 to 0.36], Standard Error of Mean 0.17
Statistical Analysis 2: Comparison: Placebo vs Naproxen; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; LS Mean Difference (Naproxen-Placebo) = -0.20, 90% CI 2-sided [-0.48 to 0.07], Standard Error of Mean 0.17
Statistical Analysis 3: Comparison: PF-06372865 vs Naproxen; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; LS Mean Difference(PF-06372865-Naproxen) = 0.28, 90% CI 2-sided [0.01 to 0.56], Standard Error of Mean 0.17
Statistical Analysis 4: Comparison: Placebo vs PF-06372865; Week 2: The mixed effect repeated measures model was used and included treatment, week, baseline, the week * treatment interaction, and the baseline * week interaction as fixed effects and week repeated within each participant as a repeated effect. Baseline was included as a covariate; Test type: Superiority or Other; LS Mean Difference (PF-06372865-Placebo) = -0.05, 90% CI 2-sided [-0.43 to 0.34], Standard Error of Mean 0.24
Statistical Analysis 5: Comparison: Placebo vs Naproxen; [analysis description as in outcome 8, analysis 4]; Test type: Superiority or Other; LS Mean Difference (Naproxen-Placebo) = -0.24, 90% CI 2-sided [-0.62 to 0.15], Standard Error of Mean 0.23
Statistical Analysis 6: Comparison: PF-06372865 vs Naproxen; [analysis description as in outcome 8, analysis 4]; Test type: Superiority or Other; LS Mean Difference(PF-06372865-Naproxen) = 0.19, 90% CI 2-sided [-0.19 to 0.58], Standard Error of Mean 0.23
Statistical Analysis 7: Comparison: Placebo vs PF-06372865; Week 3: The mixed effect repeated measures model was used and included treatment, week, baseline, the week * treatment interaction, and the baseline * week interaction as fixed effects and week repeated within each participant as a repeated effect. Baseline was included as a covariate; Test type: Superiority or Other; LS Mean Difference (PF-06372865-Placebo) = 0.03, 90% CI 2-sided [-0.39 to 0.45], Standard Error of Mean 0.26
Statistical Analysis 8: Comparison: Placebo vs Naproxen; [analysis description as in outcome 8, analysis 7]; Test type: Superiority or Other; LS Mean Difference (Naproxen-Placebo) = -0.27, 90% CI 2-sided [-0.69 to 0.16], Standard Error of Mean 0.26
Statistical Analysis 9: Comparison: PF-06372865 vs Naproxen; [analysis description as in outcome 8, analysis 7]; Test type: Superiority or Other; LS Mean Difference(PF-06372865-Naproxen) = 0.30, 90% CI [-0.12 to 0.71], Standard Error of Mean 0.25
Statistical Analysis 10: Comparison: Placebo vs PF-06372865; Week 4: The mixed effect repeated measures model was used and included treatment, week, baseline, the week * treatment interaction, and the baseline * week interaction as fixed effects and week repeated within each participant as a repeated effect. Baseline was included as a covariate; Test type: Superiority or Other; LS Mean Difference (PF-06372865-Placebo) = 0.07, 90% CI 2-sided [-0.40 to 0.55], Standard Error of Mean 0.29
Statistical Analysis 11: Comparison: Placebo vs Naproxen; [analysis description as in outcome 8, analysis 10]; Test type: Superiority or Other; LS Mean Difference (Naproxen-Placebo) = -0.37, 90% CI 2-sided [-0.84 to 0.11], Standard Error of Mean 0.29
Statistical Analysis 12: Comparison: PF-06372865 vs Naproxen; [analysis description as in outcome 8, analysis 10]; Test type: Superiority or Other; LS Mean Difference(PF-06372865-Naproxen) = 0.44, 90% CI 2-sided [-0.03 to 0.91], Standard Error of Mean 0.28

9. Secondary Outcome: Percent Change From Baseline in Daily Low Back Pain Intensity (LBPI) as Measured by an 11-point Numeric Rating Scale (NRS) at Week 1, 2, 3 and 4
Description: as for outcome 8
Time Frame: Baseline, Week 1, 2, 3, 4
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-06372865 | Naproxen
Number analyzed (Participants) | 74 | 74 | 74
percent change
  Change at week 1 (n= 74, 74, 74) | -7.453 (18.2639) [0.87 to 0.94] | -5.830 (16.0979) [0.89 to 0.97] | -10.601 (17.4139) [0.84 to 0.91]
  Change at week 2 (n= 65, 70, 72) | -15.190 (21.7655) [0.76 to 0.87] | -15.467 (20.4505) [0.77 to 0.88] | -17.682 (24.3704) [0.73 to 0.83]
  Change at week 3 (n= 62, 69, 70) | -19.100 (25.5461) | -17.167 (23.7288) | -22.204 (23.2540)
  Change at week 4 (n= 59, 64, 66) | -20.958 (25.5848) | -17.072 (27.4016) | -23.906 (28.0190)
Statistical Analysis 1: Comparison: Placebo vs PF-06372865; Week 1: The mixed effect repeated measures model includes treatment, week and the week*treatment interaction as fixed effects, week repeated within each subject as a repeated effect and log baseline as a response. LS Mean Difference and 90 percent confidence interval was calculated from log values; Test type: Superiority or Other; LS Mean Difference (PF-06372865-Placebo) = 0.03, 90% CI 2-sided [-0.03 to 0.08], Standard Error of Mean 0.03
Statistical Analysis 2: Comparison: Placebo vs Naproxen; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; LS Mean Difference (Naproxen-Placebo) = -0.04, 90% CI 2-sided [-0.09 to 0.02], Standard Error of Mean 0.03
Statistical Analysis 3: Comparison: PF-06372865 vs Naproxen; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; LS Mean Difference(PF-06372865-Naproxen) = 0.06, 90% CI 2-sided [0.01 to 0.12], Standard Error of Mean 0.03
Statistical Analysis 4: Comparison: Placebo vs PF-06372865; Week 2: The mixed effect repeated measures model includes treatment, week and the week*treatment interaction as fixed effects, week repeated within each subject as a repeated effect and log baseline as a response. LS Mean Difference and 90 percent confidence interval was calculated from log values; Test type: Superiority or Other; LS Mean Difference (PF-06372865-Placebo) = 0.01, 90% CI 2-sided [-0.09 to 0.10], Standard Error of Mean 0.06
Statistical Analysis 5: Comparison: Placebo vs Naproxen; [analysis description as in outcome 9, analysis 4]; Test type: Superiority or Other; LS Mean Difference (Naproxen-Placebo) = -0.05, 90% CI 2-sided [-0.15 to 0.05], Standard Error of Mean 0.06
Statistical Analysis 6: Comparison: PF-06372865 vs Naproxen; [analysis description as in outcome 9, analysis 4]; Test type: Superiority or Other; LS Mean Difference(PF-06372865-Naproxen) = 0.06, 90% CI 2-sided [-0.04 to 0.15], Standard Error of Mean 0.06
Statistical Analysis 7: Comparison: Placebo vs PF-06372865; Week 3: The mixed effect repeated measures model includes treatment, week and the week*treatment interaction as fixed effects, week repeated within each subject as a repeated effect and log baseline as a response. LS Mean Difference and 90 percent confidence interval was calculated from log values; Test type: Superiority or Other; LS Mean Difference (PF-06372865-Placebo) = 0.00, 90% CI 2-sided [-0.12 to 0.12], Standard Error of Mean 0.07
Statistical Analysis 8: Comparison: Placebo vs Naproxen; [analysis description as in outcome 9, analysis 7]; Test type: Superiority or Other; LS Mean Difference (Naproxen-Placebo) = -0.05, 90% CI 2-sided [-0.16 to 0.07], Standard Error of Mean 0.07
Statistical Analysis 9: Comparison: PF-06372865 vs Naproxen; [analysis description as in outcome 9, analysis 7]; Test type: Superiority or Other; LS Mean Difference(PF-06372865-Naproxen) = 0.05, 90% CI 2-sided [-0.07 to 0.16], Standard Error of Mean 0.07
Statistical Analysis 10: Comparison: Placebo vs PF-06372865; Week 4: The mixed effect repeated measures model includes treatment, week and the week*treatment interaction as fixed effects, week repeated within each subject as a repeated effect and log baseline as a response. LS Mean Difference and 90 percent confidence interval was calculated from log values; Test type: Superiority or Other; LS Mean Difference (PF-06372865-Placebo) = -0.01, 90% CI 2-sided [-0.16 to 0.14], Standard Error of Mean 0.09
Statistical Analysis 11: Comparison: Placebo vs Naproxen; [analysis description as in outcome 9, analysis 10]; Test type: Superiority or Other; LS Mean Difference (Naproxen-Placebo) = -0.10, 90% CI 2-sided [-0.24 to 0.05], Standard Error of Mean 0.09
Statistical Analysis 12: Comparison: PF-06372865 vs Naproxen; [analysis description as in outcome 9, analysis 10]; Test type: Superiority or Other; LS Mean Difference(PF-06372865-Naproxen) = 0.09, 90% CI 2-sided [-0.05 to 0.23], Standard Error of Mean 0.09

10. Secondary Outcome: Number of Participants With Sustained Response Rates in Daily Average LBPI NRS Scores at Greater Than or Equal to (>=) 30 Percent and >=50 Percent Reduction From Baseline
Description: Average back pain was assessed with an 11-point NRS ranging from 0 (no pain) to 10 (worst possible pain), where higher scores indicated higher pain. Participants described their average low back pain during the past 24 hours by choosing the appropriate number from 0 to 10. Percentage of reduction from baseline in the daily average LBPI NRS score was calculated as: ([daily value - baseline value] divided by baseline value) multiplied by 100. Number of participants with sustained response rates (for a minimum of 4 consecutive days) in the daily average LBPI NRS scores that were at >=30 percent and >=50 percent reduced from baseline were reported.
Time Frame: Baseline up to Week 4
Population: FAS included all participants randomized and who had received at least 1 dose of randomized treatment.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-06372865 | Naproxen
Number analyzed (Participants) | 74 | 74 | 74
participants
  >=30 percent response | 25 (1.351) [-1.50 to -0.89] | 24 (1.091) [-1.35 to -0.71] | 31 (1.401) [-1.77 to -1.14]
  >=50 percent response | 11 | 9 | 12
Statistical Analysis 1: Comparison: Placebo vs PF-06372865; >=30 percent sustained response rates: Odds Ratios based on a logistic regression model included treatment as a fixed effect and baseline as a covariate; Test type: Superiority or Other; Odds Ratio (OR) = 0.97, 90% CI 2-sided [0.54 to 1.73]
Statistical Analysis 2: Comparison: Placebo vs Naproxen; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; Odds Ratio (OR) = 1.43, 90% CI 2-sided [0.81 to 2.51]
Statistical Analysis 3: Comparison: PF-06372865 vs Naproxen; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; Odds Ratio (OR) = 0.68, 90% CI 2-sided [0.39 to 1.20]
Statistical Analysis 4: Comparison: Placebo vs PF-06372865; >=50 percent sustained response rates: Odds Ratios based on a logistic regression model included treatment as a fixed effect and baseline as a covariate; Test type: Superiority or Other; Odds Ratio (OR) = 0.81, 90% CI 2-sided [0.37 to 1.81]
Statistical Analysis 5: Comparison: Placebo vs Naproxen; [analysis description as in outcome 10, analysis 4]; Test type: Superiority or Other; Odds Ratio (OR) = 1.11, 90% CI 2-sided [0.53 to 2.35]
Statistical Analysis 6: Comparison: PF-06372865 vs Naproxen; [analysis description as in outcome 10, analysis 4]; Test type: Superiority or Other; Odds Ratio (OR) = 0.73, 90% CI 2-sided [0.33 to 1.60]

11. Secondary Outcome: Number of Participants Withdrawn Due to Lack of Efficacy
Description: Participants withdrew from the study due to lack of efficacy (insufficient clinical response) were reported.
Time Frame: Baseline up to Week 4
Population: FAS included all participants randomized and who had received at least 1 dose of randomized treatment.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-06372865 | Naproxen
Number analyzed (Participants) | 74 | 74 | 74
participants | 2 (1.351) [-1.50 to -0.89] | 0 (1.091) [-1.35 to -0.71] | 1 (1.401) [-1.77 to -1.14]

12. Secondary Outcome: Time to Withdrawal Due to Lack of Efficacy
Description: Kaplan Meier and Cox Proportional Hazards analyses were to be used to compute the time to withdrawal due to lack of efficacy. Withdrawal due to lack of efficacy was identified from the participant summary case report form (CRF) page and where reason was identified as "Insufficient Clinical Response". Time to withdrawal was calculated as Date of withdrawal - Date of Randomization.
Time Frame: Baseline up to Week 4
Population: FAS included all participants randomized and who had received at least 1 dose of randomized treatment.
Measure: Median (90% Confidence Interval); unit: days
Arm/Group | Placebo | PF-06372865 | Naproxen
Number analyzed (Participants) | 74 | 74 | 74
days | NA (1.351) [NA to NA] — Outcome was to be assessed as time to event analysis by Kaplan-Meier estimates. However, median and 90% CI were not estimable since very few participants withdrew from study due to lack of efficacy: 2 in placebo group, 1 in naproxen group. | NA (1.091) [NA to NA] — Outcome was to be assessed as time to event analysis by Kaplan-Meier estimates. However, median and 90% CI were not estimable since very few participants withdrew from study due to lack of efficacy: 2 in placebo group, 1 in naproxen group. | NA (1.401) [NA to NA] — Outcome was to be assessed as time to event analysis by Kaplan-Meier estimates. However, median and 90% CI were not estimable since very few participants withdrew from study due to lack of efficacy: 2 in placebo group, 1 in naproxen group.

13. Secondary Outcome: Number of Participants Using Rescue Medication
Description: Participants were permitted to use any commercial product (tablet/caplet/capsule) of acetaminophen (paracetamol) 500 mg as a rescue medication. Number of participants who used rescue medication were reported.
Time Frame: Week 1, 2, 3, 4
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Placebo | PF-06372865 | Naproxen
Number analyzed (Participants) | 74 | 74 | 74
participants
  Week 1 (n= 74, 74, 74) | 34 (1.351) [-1.50 to -0.89] | 35 (1.091) [-1.35 to -0.71] | 34 (1.401) [-1.77 to -1.14]
  Week 2 (n= 67, 72, 72) | 26 | 32 | 30
  Week 3 (n= 63, 69, 71) | 25 | 31 | 27
  Week 4 (59, 66, 67) | 23 | 27 | 22

14. Secondary Outcome: Number of Days Participants Used the Rescue Medication
Description: The number of days for which the participants used the rescue medication were reported. Participants recorded the usage of acetaminophen rescue medication in the daily diary.
Time Frame: Week 1, 2, 3, 4
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | PF-06372865 | Naproxen
Number analyzed (Participants) | 74 | 74 | 74
days
  Week 1 (n= 74, 74, 74) | 1.7 (2.62) [-1.50 to -0.89] | 1.7 (2.49) [-1.35 to -0.71] | 1.7 (2.44) [-1.77 to -1.14]
  Week 2 (n= 67, 72, 72) | 1.6 (2.65) | 1.8 (2.77) | 1.6 (2.54)
  Week 3 (n= 63, 69, 71) | 1.9 (3.11) | 1.4 (2.22) | 1.5 (2.46)
  Week 4 (59, 66, 67) | 1.4 (2.37) | 1.4 (2.15) | 1.4 (2.45)

15. Secondary Outcome: Amount of Rescue Medication Used by the Participants
Description: The amount of rescue medication (Acetaminophen [paracetamol]) used was reported. Participants were permitted to use any commercial product of acetaminophen tablet/caplet/capsule.
Time Frame: Week 1, 2, 3, 4
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Placebo | PF-06372865 | Naproxen
Number analyzed (Participants) | 74 | 74 | 74
mg
  Week 1 (n= 72, 70, 74) | 1388.9 (2703.97) [-1.50 to -0.89] | 1621.8 (4169.38) [-1.35 to -0.71] | 2064.5 (4298.80) [-1.77 to -1.14]
  Week 2 (n= 65, 68, 72) | 1030.8 (1669.76) | 1594.1 (3708.11) | 1920.5 (4327.48)
  Week 3 (n= 61, 65, 71) | 1172.1 (1955.52) | 1416.9 (3552.05) | 1740.5 (4361.26)
  Week 4 (n= 58, 62, 67) | 1101.7 (2069.03) | 1348.8 (2925.65) | 1489.2 (3567.20)

16. Secondary Outcome: Change From Baseline in Roland-Morris Disability Questionnaire (RMDQ) Total Score at Week 1, 2, and 3
Description: Each participant assessed his or her own disability due to low back pain using the RMDQ worksheet. The RMDQ total score was calculated as the total number of statements that were checked; the RMDQ total possible scores ranges from 0 to 24, with higher scores indicating greater disability.
Time Frame: Baseline, Week 1, 2, 3
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | PF-06372865 | Naproxen
Number analyzed (Participants) | 74 | 74 | 74
units on a scale
  Baseline (n= 74, 74, 74) | 9.8 (5.47) | 9.4 (5.23) | 8.5 (5.48)
  Change at week 1 (n= 73, 73, 73) | -0.4 (2.48) | -0.5 (3.73) | -1.2 (3.51)
  Change at week 2 (n= 66, 71, 72) | -0.7 (3.17) | -1.3 (3.59) | -1.6 (4.07)
  Change at week 3 (n= 62, 67, 71) | -1.0 (3.24) | -1.3 (3.39) | -2.0 (4.21)
Statistical Analysis 1: Comparison: Placebo vs PF-06372865; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; LS Mean Difference (PF-06372865-Placebo) = -0.18, 90% CI 2-sided [-1.06 to 0.70], Standard Error of Mean 0.53
Statistical Analysis 2: Comparison: Placebo vs Naproxen; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; LS Mean Difference (Naproxen-Placebo) = -0.91, 90% CI 2-sided [-1.80 to -0.03], Standard Error of Mean 0.53
Statistical Analysis 3: Comparison: PF-06372865 vs Naproxen; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; LS Mean Difference(PF-06372865-Naproxen) = 0.73, 90% CI 2-sided [-0.15 to 1.61], Standard Error of Mean 0.53
Statistical Analysis 4: Comparison: Placebo vs PF-06372865; [analysis description as in outcome 8, analysis 4]; Test type: Superiority or Other; LS Mean Difference (PF-06372865-Placebo) = -0.70, 90% CI 2-sided [-1.69 to 0.29], Standard Error of Mean 0.60
Statistical Analysis 5: Comparison: Placebo vs Naproxen; [analysis description as in outcome 8, analysis 4]; Test type: Superiority or Other; LS Mean Difference (Naproxen-Placebo) = -1.11, 90% CI 2-sided [-2.11 to -0.11], Standard Error of Mean 0.60
Statistical Analysis 6: Comparison: PF-06372865 vs Naproxen; [analysis description as in outcome 8, analysis 4]; Test type: Superiority or Other; LS Mean Difference(PF-06372865-Naproxen) = 0.41, 90% CI 2-sided [-0.57 to 1.39], Standard Error of Mean 0.59
Statistical Analysis 7: Comparison: Placebo vs PF-06372865; [analysis description as in outcome 8, analysis 7]; Test type: Superiority or Other; LS Mean Difference (PF-06372865-Placebo) = -0.41, 90% CI 2-sided [-1.42 to 0.60], Standard Error of Mean 0.61
Statistical Analysis 8: Comparison: Placebo vs Naproxen; [analysis description as in outcome 8, analysis 7]; Test type: Superiority or Other; LS Mean Difference (Naproxen-Placebo) = -1.27, 90% CI 2-sided [-2.28 to -0.27], Standard Error of Mean 0.61
Statistical Analysis 9: Comparison: PF-06372865 vs Naproxen; [analysis description as in outcome 8, analysis 7]; Test type: Superiority or Other; LS Mean Difference(PF-06372865-Naproxen) = 0.86, 90% CI 2-sided [-0.12 to 1.85], Standard Error of Mean 0.60

17. Secondary Outcome: Change From Baseline in Roland-Morris Disability Questionnaire (RMDQ) Total Score at Week 4
Description: as for outcome 16
Time Frame: Baseline, Week 4
Population: FAS included all participants randomized and who had received at least 1 dose of randomized treatment.
Measure: Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | PF-06372865 | Naproxen
Number analyzed (Participants) | 74 | 74 | 74
units on a scale | -1.00 (3.36) [-1.67 to -0.33] | -1.64 (3.85) [-2.35 to -0.92] | -2.43 (4.73) [-3.14 to -1.71]
Statistical Analysis 1: Comparison: Placebo vs PF-06372865; Week 4: An ANCOVA model within an outlier robust Bayesian framework was applied. Baseline was included as a fixed effect. An informative N (-3.28, 1.19^2) prior for the placebo effect was assumed. Non informative prior distributions were assumed for the rest of the model parameters. LOCF was used for missing data; Test type: Superiority or Other; Mean Difference (PF-06372865-Placebo) = -0.64, 90% CI 2-sided [-1.63 to 0.35]
Statistical Analysis 2: Comparison: Placebo vs Naproxen; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; Mean Difference (Naproxen-Placebo) = -1.43, 90% CI 2-sided [-2.40 to -0.45]
Statistical Analysis 3: Comparison: PF-06372865 vs Naproxen; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; Mean Difference (PF-06372865-Naproxen) = 0.79, 90% CI 2-sided [-0.22 to 1.80]

18. Secondary Outcome: Change From Baseline in Hopkins Verbal Learning Test-Revised (HVLT-R) at Week 2 and 4
Description: This test assesses verbal learning and memory. Participants are given a list of 12 words and asked to repeat as many words as they can recall during 3 separate learning trials. The total recall score ranges from 0 (no memory) to 36 (best memory) while the delayed recall trial score ranges from 0 (no memory) to 12 (best memory); higher scores indicated greater verbal learning and recall.
Time Frame: Baseline, Week 2, Week 4
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | PF-06372865 | Naproxen
Number analyzed (Participants) | 74 | 74 | 74
units on a scale
  Total recall score: at Baseline (n= 74,74,74) | 24.47 (5.118) | 22.92 (5.581) | 24.46 (5.455)
  Total recall score: Change at Week 2 (n= 66,72,71) | 0.74 (3.702) [-0.28 to 0.62] | 0.57 (3.950) [-1.03 to -0.17] | -0.30 (4.773) [-0.44 to 0.43]
  Total recall score: Change at Week 4 (n= 56,66,66) | 1.43 (3.637) [-0.03 to 1.62] | 0.68 (3.522) | 0.11 (4.062)
  Delayed Recall Score: at Baseline (n= 74,74,74) | 8.59 (2.415) | 8.31 (2.828) | 8.59 (2.643)
  Delayed Recall Score:Change at Week 2 (n=66,72,71) | 0.18 (2.225) | -0.57 (2.803) | -0.06 (1.912)
  Delayed Recall Score:Change at Week 4 (n=56,65,66) | 0.57 (1.925) | -0.28 (2.197) | 0.41 (1.831)
Statistical Analysis 1: Comparison: Placebo vs PF-06372865; Total recall score at Week 2: The mixed effect repeated measures model was used and included treatment, week, baseline, the week * treatment interaction, and the baseline * week interaction as fixed effects and week repeated within each participant as a repeated effect. Baseline (recordings on Day 1) was included as a covariate. Unplanned readings were excluded from the analysis; Test type: Superiority or Other; LS Mean Difference (PF-06372865-Placebo) = -0.37, 90% CI 2-sided [-1.52 to 0.78], Standard Error of Mean 0.70
Statistical Analysis 2: Comparison: Placebo vs Naproxen; [analysis description as in outcome 18, analysis 1]; Test type: Superiority or Other; LS Mean Difference (Naproxen-Placebo) = -0.95, 90% CI 2-sided [-2.10 to 0.20], Standard Error of Mean 0.70
Statistical Analysis 3: Comparison: PF-06372865 vs Naproxen; [analysis description as in outcome 18, analysis 1]; Test type: Superiority or Other; LS Mean Difference(PF-06372865-Naproxen) = 0.58, 90% CI 2-sided [-0.56 to 1.71], Standard Error of Mean 0.68
Statistical Analysis 4: Comparison: Placebo vs PF-06372865; Total Recall score at Week 4: The mixed effect repeated measures model was used and included treatment, week, baseline, the week * treatment interaction, and the baseline * week interaction as fixed effects and week repeated within each participant as a repeated effect. Baseline (recordings on Day 1) was included as a covariate. Unplanned readings were excluded from the analysis; Test type: Superiority or Other; LS Mean Difference (PF-06372865-Placebo) = -1.02, 90% CI 2-sided [-2.06 to 0.02], Standard Error of Mean 0.63
Statistical Analysis 5: Comparison: Placebo vs Naproxen; [analysis description as in outcome 18, analysis 4]; Test type: Superiority or Other; LS Mean Difference (Naproxen-Placebo) = -1.21, 90% CI 2-sided [-2.25 to -0.17], Standard Error of Mean 0.63
Statistical Analysis 6: Comparison: PF-06372865 vs Naproxen; [analysis description as in outcome 18, analysis 4]; Test type: Superiority or Other; LS Mean Difference(PF-06372865-Naproxen) = 0.19, 90% CI 2-sided [-0.82 to 1.19], Standard Error of Mean 0.61
Statistical Analysis 7: Comparison: Placebo vs PF-06372865; Delayed recall score at Week 2: The mixed effect repeated measures model was used and included treatment, week, baseline, the week * treatment interaction, and the baseline * week interaction as fixed effects and week repeated within each participant as a repeated effect. Baseline (recordings on Day 1) was included as a covariate. Unplanned readings were excluded from the analysis; Test type: Superiority or Other; LS Mean Difference (PF-06372865-Placebo) = -0.77, 90% CI 2-sided [-1.39 to -0.15], Standard Error of Mean 0.38
Statistical Analysis 8: Comparison: Placebo vs Naproxen; [analysis description as in outcome 18, analysis 7]; Test type: Superiority or Other; LS Mean Difference (Naproxen-Placebo) = -0.17, 90% CI 2-sided [-0.80 to 0.45], Standard Error of Mean 0.38
Statistical Analysis 9: Comparison: PF-06372865 vs Naproxen; [analysis description as in outcome 18, analysis 7]; Test type: Superiority or Other; LS Mean Difference(PF-06372865-Naproxen) = -0.60, 90% CI 2-sided [-1.21 to 0.02], Standard Error of Mean 0.37
Statistical Analysis 10: Comparison: Placebo vs PF-06372865; Delayed recall score at Week 4: The mixed effect repeated measures model was used and included treatment, week, baseline, the week * treatment interaction, and the baseline * week interaction as fixed effects and week repeated within each participant as a repeated effect. Baseline (recordings on Day 1) was included as a covariate. Unplanned readings were excluded from the analysis; Test type: Superiority or Other; LS Mean Difference (PF-06372865-Placebo) = -0.85, 90% CI 2-sided [-1.42 to -0.28], Standard Error of Mean 0.34
Statistical Analysis 11: Comparison: Placebo vs Naproxen; [analysis description as in outcome 18, analysis 10]; Test type: Superiority or Other; LS Mean Difference (Naproxen-Placebo) = -0.11, 90% CI 2-sided [-0.67 to 0.46], Standard Error of Mean 0.34
Statistical Analysis 12: Comparison: PF-06372865 vs Naproxen; [analysis description as in outcome 18, analysis 10]; Test type: Superiority or Other; LS Mean Difference(PF-06372865-Naproxen) = -0.74, 90% CI 2-sided [-1.29 to -0.20], Standard Error of Mean 0.33

19. Secondary Outcome: Chronic Low Back Pain (CLBP) Responder Index Analysis
Description: Participants were successful responders if they had any of the following: >=30 percent reduction in mean daily average LBPI from baseline to particular week; decrease of >=30 percent in participant's global assessment of low back pain (disease activity) from baseline to particular week or no worsening (increase) in RMDQ total score from baseline to particular week.
Time Frame: Week 1, 2, 3, 4
Population: FAS included all participants randomized and who had received at least 1 dose of randomized treatment.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-06372865 | Naproxen
Number analyzed (Participants) | 74 | 74 | 74
participants
  Week 1 | 0 (2.62) [-1.50 to -0.89] | 0 (2.49) [-1.35 to -0.71] | 8 (2.44) [-1.77 to -1.14]
  Week 2 | 5 (2.65) | 8 (2.77) | 11 (2.54)
  Week 3 | 12 (3.11) | 8 (2.22) | 14 (2.46)
  Week 4 | 9 (2.37) | 11 (2.15) | 19 (2.45)
Statistical Analysis 1: Comparison: Placebo vs PF-06372865; A repeated measures logistic regression model included treatment and week as fixed effects and LBPI baseline as a covariate. Participant was included as a repeated effect; Test type: Superiority or Other; Odds Ratio (OR) = 0.98, 90% CI 2-sided [0.61 to 1.58]
Statistical Analysis 2: Comparison: Placebo vs Naproxen; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; Odds Ratio (OR) = 2.04, 90% CI 2-sided [1.33 to 3.14]
Statistical Analysis 3: Comparison: PF-06372865 vs Naproxen; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; Odds Ratio (OR) = 0.48, 90% CI 2-sided [0.31 to 0.74]

20. Secondary Outcome: Change From Baseline in Participant's Global Assessment (PtGA) of Low Back Pain Score at Week 1, 2, 3 and 4
Description: Participant rated 5-point Likert scale ranging from 0 (no pain) to 4 (worst possible pain) with a higher score indicating greater level of pain.
Time Frame: Baseline, Week 1, 2, 3, 4
Population: as for outcome 8
Measure: Least Squares Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | PF-06372865 | Naproxen
Number analyzed (Participants) | 74 | 74 | 74
units on a scale
  Change at Week 1 (n= 73, 73, 73) | -0.20 [-0.33 to -0.06] | -0.19 [-0.33 to -0.05] | -0.34 [-0.48 to -0.20]
  Change at Week 2 (n= 66, 71, 72) | -0.24 [-0.40 to -0.09] | -0.28 [-0.43 to -0.13] | -0.39 [-0.55 to -0.24]
  Change at Week 3 (n= 62, 67, 71) | -0.45 [-0.62 to -0.29] | -0.31 [-0.47 to -0.14] | -0.43 [-0.60 to -0.27]
  Change at Week 4 (n= 58, 65, 65) | -0.33 [-0.52 to -0.15] | -0.21 [-0.38 to -0.03] | -0.54 [-0.71 to -0.36]
Statistical Analysis 1: Comparison: Placebo vs PF-06372865; Week 1: The mixed effect repeated measures model was used and included treatment, week, baseline, the week * treatment interaction, and the baseline * week interaction as fixed effects and week repeated within each participant as a repeated effect. Baseline (recordings on Day 1) was included as a covariate; Test type: Superiority or Other; LS Mean Difference (PF-06372865-Placebo) = 0.01, 90% CI 2-sided [-0.19 to 0.20], Standard Error of Mean 0.12
Statistical Analysis 2: Comparison: Placebo vs Naproxen; [analysis description as in outcome 20, analysis 1]; Test type: Superiority or Other; LS Mean Difference (Naproxen-Placebo) = -0.14, 90% CI 2-sided [-0.34 to 0.05], Standard Error of Mean 0.12
Statistical Analysis 3: Comparison: PF-06372865 vs Naproxen; [analysis description as in outcome 20, analysis 1]; Test type: Superiority or Other; LS Mean Difference(PF-06372865-Naproxen) = 0.15, 90% CI 2-sided [-0.05 to 0.35], Standard Error of Mean 0.12
Statistical Analysis 4: Comparison: Placebo vs PF-06372865; Week 2: The mixed effect repeated measures model was used and included treatment, week, baseline, the week * treatment interaction, and the baseline * week interaction as fixed effects and week repeated within each participant as a repeated effect. Baseline (recordings on Day 1) was included as a covariate; Test type: Superiority or Other; LS Mean Difference (PF-06372865-Placebo) = -0.04, 90% CI 2-sided [-0.26 to 0.18], Standard Error of Mean 0.13
Statistical Analysis 5: Comparison: Placebo vs Naproxen; [analysis description as in outcome 20, analysis 4]; Test type: Superiority or Other; LS Mean Difference (Naproxen-Placebo) = -0.15, 90% CI 2-sided [-0.37 to 0.07], Standard Error of Mean 0.13
Statistical Analysis 6: Comparison: PF-06372865 vs Naproxen; [analysis description as in outcome 20, analysis 4]; Test type: Superiority or Other; LS Mean Difference(PF-06372865-Naproxen) = 0.11, 90% CI 2-sided [-0.10 to 0.33], Standard Error of Mean 0.13
Statistical Analysis 7: Comparison: Placebo vs PF-06372865; Week 3: The mixed effect repeated measures model was used and included treatment, week, baseline, the week * treatment interaction, and the baseline * week interaction as fixed effects and week repeated within each participant as a repeated effect. Baseline (recordings on Day 1) was included as a covariate; Test type: Superiority or Other; LS Mean Difference (PF-06372865-Placebo) = 0.15, 90% CI 2-sided [-0.09 to 0.38], Standard Error of Mean 0.14
Statistical Analysis 8: Comparison: Placebo vs Naproxen; [analysis description as in outcome 20, analysis 7]; Test type: Superiority or Other; LS Mean Difference (Naproxen-Placebo) = 0.02, 90% CI 2-sided [-0.21 to 0.25], Standard Error of Mean 0.14
Statistical Analysis 9: Comparison: PF-06372865 vs Naproxen; [analysis description as in outcome 20, analysis 7]; Test type: Superiority or Other; LS Mean Difference(PF-06372865-Naproxen) = 0.13, 90% CI 2-sided [-0.10 to 0.36], Standard Error of Mean 0.14
Statistical Analysis 10: Comparison: Placebo vs PF-06372865; Week 4: The mixed effect repeated measures model was used and included treatment, week, baseline, the week * treatment interaction, and the baseline * week interaction as fixed effects and week repeated within each participant as a repeated effect. Baseline (recordings on Day 1) was included as a covariate; Test type: Superiority or Other; LS Mean Difference (PF-06372865-Placebo) = 0.12, 90% CI 2-sided [-0.13 to 0.38], Standard Error of Mean 0.15
Statistical Analysis 11: Comparison: Placebo vs Naproxen; [analysis description as in outcome 20, analysis 10]; Test type: Superiority or Other; LS Mean Difference (Naproxen-Placebo) = -0.21, 90% CI 2-sided [-0.46 to 0.05], Standard Error of Mean 0.15
Statistical Analysis 12: Comparison: PF-06372865 vs Naproxen; [analysis description as in outcome 20, analysis 10]; Test type: Superiority or Other; LS Mean Difference(PF-06372865-Naproxen) = 0.33, 90% CI 2-sided [0.08 to 0.58], Standard Error of Mean 0.15

21. Secondary Outcome: Patient Global Impression of Change (PGI-C) Score
Description: PGI-C was a participant rated instrument to measure participant's assessment of change in his or her overall status since the previous visit on a 7-point scale; ranging from 1 (very much improved) to 7 (very much worse), where higher scores indicated more worsening.
Time Frame: Week 1, 2, 3, 4
Population: as for outcome 8
Measure: Least Squares Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | PF-06372865 | Naproxen
Number analyzed (Participants) | 74 | 74 | 74
units on a scale
  Week 1 (n= 73, 73, 73) | 3.32 [3.14 to 3.49] | 3.15 [2.97 to 3.32] | 2.95 [2.77 to 3.12]
  Week 2 (n= 66, 71, 72) | 3.12 [2.91 to 3.33] | 3.04 [2.83 to 3.24] | 2.83 [2.63 to 3.04]
  Week 3 (n= 62, 67, 71) | 3.01 [2.81 to 3.22] | 2.94 [2.74 to 3.14] | 2.63 [2.43 to 2.83]
  Week 4 (n= 58, 65, 65) | 3.04 [2.81 to 3.27] | 2.93 [2.72 to 3.15] | 2.61 [2.39 to 2.82]
Statistical Analysis 1: Comparison: Placebo vs PF-06372865; Week 1: The mixed effect repeated measures model was used and included treatment, week, baseline, the week * treatment interaction, and the baseline * week interaction as fixed effects and week repeated within each participant as a repeated effect; Test type: Superiority or Other; LS Mean Difference (PF-06372865-Placebo) = -0.17, 90% CI 2-sided [-0.42 to 0.08], Standard Error of Mean 0.15
Statistical Analysis 2: Comparison: Placebo vs Naproxen; [analysis description as in outcome 21, analysis 1]; Test type: Superiority or Other; LS Mean Difference (Naproxen-Placebo) = -0.37, 90% CI 2-sided [-0.62 to -0.12], Standard Error of Mean 0.15
Statistical Analysis 3: Comparison: PF-06372865 vs Naproxen; [analysis description as in outcome 21, analysis 1]; Test type: Superiority or Other; LS Mean Difference(PF-06372865-Naproxen) = 0.20, 90% CI 2-sided [-0.05 to 0.45], Standard Error of Mean 0.15
Statistical Analysis 4: Comparison: Placebo vs PF-06372865; Week 2: The mixed effect repeated measures model was used and included treatment, week, baseline, the week * treatment interaction, and the baseline * week interaction as fixed effects and week repeated within each participant as a repeated effect; Test type: Superiority or Other; LS Mean Difference (PF-06372865-Placebo) = -0.08, 90% CI 2-sided [-0.38 to 0.21], Standard Error of Mean 0.18
Statistical Analysis 5: Comparison: Placebo vs Naproxen; [analysis description as in outcome 21, analysis 4]; Test type: Superiority or Other; LS Mean Difference (Naproxen-Placebo) = -0.29, 90% CI 2-sided [-0.58 to 0.01], Standard Error of Mean 0.18
Statistical Analysis 6: Comparison: PF-06372865 vs Naproxen; [analysis description as in outcome 21, analysis 4]; Test type: Superiority or Other; LS Mean Difference(PF-06372865-Naproxen) = 0.20, 90% CI 2-sided [-0.09 to 0.49], Standard Error of Mean 0.18
Statistical Analysis 7: Comparison: Placebo vs PF-06372865; Week 3: The mixed effect repeated measures model was used and included treatment, week, baseline, the week * treatment interaction, and the baseline * week interaction as fixed effects and week repeated within each participant as a repeated effect; Test type: Superiority or Other; LS Mean Difference (PF-06372865-Placebo) = -0.07, 90% CI 2-sided [-0.36 to 0.21], Standard Error of Mean 0.17
Statistical Analysis 8: Comparison: Placebo vs Naproxen; [analysis description as in outcome 21, analysis 7]; Test type: Superiority or Other; LS Mean Difference (Naproxen-Placebo) = -0.38, 90% CI 2-sided [-0.67 to -0.10], Standard Error of Mean 0.17
Statistical Analysis 9: Comparison: PF-06372865 vs Naproxen; [analysis description as in outcome 21, analysis 7]; Test type: Superiority or Other; LS Mean Difference(PF-06372865-Naproxen) = 0.31, 90% CI 2-sided [0.03 to 0.59], Standard Error of Mean 0.17
Statistical Analysis 10: Comparison: Placebo vs PF-06372865; Week 4: The mixed effect repeated measures model was used and included treatment, week, baseline, the week * treatment interaction, and the baseline * week interaction as fixed effects and week repeated within each participant as a repeated effect; Test type: Superiority or Other; LS Mean Difference (PF-06372865-Placebo) = -0.11, 90% CI 2-sided [-0.42 to 0.21], Standard Error of Mean 0.19
Statistical Analysis 11: Comparison: Placebo vs Naproxen; [analysis description as in outcome 21, analysis 10]; Test type: Superiority or Other; LS Mean Difference (Naproxen-Placebo) = -0.43, 90% CI 2-sided [-0.75 to -0.12], Standard Error of Mean 0.19
Statistical Analysis 12: Comparison: PF-06372865 vs Naproxen; [analysis description as in outcome 21, analysis 10]; Test type: Superiority or Other; LS Mean Difference(PF-06372865-Naproxen) = 0.33, 90% CI 2-sided [0.02 to 0.63], Standard Error of Mean 0.19

22. Secondary Outcome: Number of Participants With Global Evaluation of Study Medication (GESM) at Week 4
Description: Participants rated their study treatment by GESM questionnaire. It was a qualitative measure of efficacy utilizing a 4-point Likert scale ranging from 1 (poor) to 4 (excellent), where higher score indicated a better overall response to the treatment. Number of participants who reported a particular score had been reported.
Time Frame: Week 4
Population: FAS included all participants randomized and who had received at least 1 dose of randomized treatment. Here, "number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-06372865 | Naproxen
Number analyzed (Participants) | 70 | 73 | 71
participants
  Poor | 8 (2.62) [-1.50 to -0.89] | 11 (2.49) [-1.35 to -0.71] | 5 (2.44) [-1.77 to -1.14]
  Fair | 26 (2.65) | 18 (2.77) | 14 (2.54)
  Good | 28 (3.11) | 36 (2.22) | 37 (2.46)
  Excellent | 8 (2.37) | 8 (2.15) | 15 (2.45)
Statistical Analysis 1: Comparison: Placebo vs PF-06372865; Odds Ratios were based on a logistic regression model and included treatment as a fixed effect; Test type: Superiority or Other; Odds Ratio (OR) = 0.85, 90% CI 2-sided [0.46 to 1.56]
Statistical Analysis 2: Comparison: Placebo vs Naproxen; Odds Ratios were based on a logistic regression model and included treatment as a fixed effect; Test type: Superiority or Other; Odds Ratio (OR) = 0.43, 90% CI 2-sided [0.23 to 0.81]
Statistical Analysis 3: Comparison: PF-06372865 vs Naproxen; Odds Ratios were based on a logistic regression model and included treatment as a fixed effect; Test type: Superiority or Other; Odds Ratio (OR) = 1.97, 90% CI 2-sided [1.06 to 3.65]

23. Secondary Outcome: Plasma Concentration of PF-06372865
Description: Data was calculated by setting concentration values below the lower limit of quantification (LLOQ) to zero. The LLOQ was <0.0100 nanogram per milliliter (ng/mL).
Time Frame: Baseline, Week 1, 2, 3, 4
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-06372865
Number analyzed (Participants) | 74
ng/mL
  Baseline (n= 73) | NA (NA) — Data was not collected at baseline since number of observations above lower limit of quantification (NALQ) = 0.
  Week 1 (n= 74) | 15.57 (13.214)
  Week 2 (n= 72) | 47.51 (45.668)
  Week 3 (n= 71) | 46.65 (46.305)
  Week 4 (n= 65) | 48.24 (41.975)

24. Secondary Outcome: Plasma Concentration of Naproxen
Description: Data was calculated by setting concentration values below the LLOQ to zero. The LLOQ was <1000 ng/mL.
Time Frame: Baseline, Week 1, 2, 3, 4
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Naproxen
Number analyzed (Participants) | 74
ng/mL
  Baseline (n= 73) | 317.0 (1963.4)
  Week 1 (n= 74) | 68150 (35213)
  Week 2 (n= 72) | 67830 (37004)
  Week 3 (n= 71) | 67140 (38336)
  Week 4 (n= 65) | 65650 (33419)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo | PF-06372865 | Naproxen
Serious Adverse Events (participants affected / at risk) | 1/74 | 1/74 | 2/74
Other Adverse Events (participants affected / at risk) | 25/74 | 34/74 | 26/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=74) | PF-06372865 (N=74) | Naproxen (N=74)
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Ileus paralytic (Gastrointestinal disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=74) | PF-06372865 (N=74) | Naproxen (N=74)
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 6 | 3
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 1
Eye haemorrhage (Eye disorders) | 0 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 0
Chills (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 1
Pain (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1
Ear infection (Infections and infestations) | 0 | 1 | 0
Fungal infection (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 3 | 3
Pneumonia (Infections and infestations) | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 2
Tooth infection (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 2
Incision site pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Electrocardiogram abnormal (Investigations) | 0 | 0 | 1
Intraocular pressure increased (Investigations) | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 1 | 0
Disturbance in attention (Nervous system disorders) | 1 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 6 | 0
Head discomfort (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 5 | 1 | 1
Hypersomnia (Nervous system disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Sedation (Nervous system disorders) | 0 | 2 | 0
Somnolence (Nervous system disorders) | 1 | 9 | 1
Tinel's sign (Nervous system disorders) | 0 | 1 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 1
Panic attack (Psychiatric disorders) | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 1
Acute prerenal failure (Renal and urinary disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Breast cyst (Reproductive system and breast disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.